CLINICAL TRIAL: NCT03916250
Title: A PHASE 1, SINGLE-CENTER, RANDOMIZED, VEHICLE AND WHITE PETROLATUM CONTROLLED, EVALUATOR BLINDED STUDY TO ASSESS THE SKIN IRRITATION POTENTIAL WITH A RANGE OF CONCENTRATIONS OF PF-06700841 CREAM IN ADULT JAPANESE HEALTHY PARTICIPANTS
Brief Title: Evaluation of Skin Irritation Potential With PF-06700841 Cream Formulation Using Negative Control in Adult Japanese Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: B7931029
Record Dates: First submitted 2019-03-20; First posted 2019-04-16 (Actual); Last update posted 2019-05-24 (Actual); Status verified 2019-05

CONDITIONS: Healthy
MeSH Terms: interventions — Petrolatum

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- PF-06700841 cream 0% (Experimental): All participants will have 6 application sites where 6 patches of investigational products will be completely randomly assigned, for the purpose of determining irritation potential
  Interventions: Drug: PF-06700841 cream
- PF-06700841 cream 0.1% (Experimental): All participants will have 6 application sites where 6 patches of investigational products will be completely randomly assigned, for the purpose of determining irritation potential
  Interventions: Drug: PF-06700841 cream
- PF-06700841 cream 0.3% (Experimental): All participants will have 6 application sites where 6 patches of investigational products will be completely randomly assigned, for the purpose of determining irritation potential
  Interventions: Drug: PF-06700841 cream
- PF-06700841 cream 1% (Experimental): All participants will have 6 application sites where 6 patches of investigational products will be completely randomly assigned, for the purpose of determining irritation potential
  Interventions: Drug: PF-06700841 cream
- PF-06700841 cream 3% (Experimental): All participants will have 6 application sites where 6 patches of investigational products will be completely randomly assigned, for the purpose of determining irritation potential
  Interventions: Drug: PF-06700841 cream
- White petrolatum (Experimental): All participants will have 6 application sites where 6 patches of investigational products will be completely randomly assigned, for the purpose of determining irritation potential
  Interventions: Drug: White petrolatum

INTERVENTIONS:
Drug: PF-06700841 cream — PF-06700841 will be applied topically
  Other Names: PF-06700841 cream 0% is Vehicle
  Arms: PF-06700841 cream 0%; PF-06700841 cream 0.1%; PF-06700841 cream 0.3%; PF-06700841 cream 1%; PF-06700841 cream 3%
Drug: White petrolatum — White petrolatum will be applied topically
  Arms: White petrolatum

SUMMARY:
This is a Phase 1, single center, randomized, vehicle and white petrolatum controlled, evaluator blinded study to assess the skin irritation potential with a range of concentrations of PF-06700841 cream including vehicle and empty patch with white petrolatum under occlusive conditions in adult Japanese healthy participants.

ELIGIBILITY:
Inclusion Criteria:

* Male and female participants must be 20 to 55 years of age, inclusive, at the time of signing the informed consent document.
* Body mass index (BMI) of 17.5 to 25 kg/m2; and a total body weight >50 kg (110 lb).

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurological, or allergic disease.
* Participants who have any visible skin condition at the application site which, in the opinion of the investigative personnel, will interfere with the evaluation of the test site reaction.
* Participants who have psoriasis and/or active AD/eczema/urticaria.
* Participants who have a history of AD.
* Participants who have damaged skin in or around the test sites, including sunburn, excessively deep tans, uneven skin tones, tattoos, scars, excessive hair, numerous freckles, or other disfigurations of the test site.
* History of known or suspected intolerance to any of the ingredients of the investigational products, adhesive tape/plaster, or the test patches.

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2019-03-23 (Actual); Primary Completion 2019-04-15 (Actual); Study Completion 2019-05-12 (Actual)

PRIMARY OUTCOMES:
The proportion of participants who have skin irritation grade equal to or greater than two plus (++) up to Day 4 | Up to Day 4
  Skin irritation grade is defined as following: no reaction (-); slight erythema (+-); erythema (+); erythema + edema, papules (++); erythema + edema + papules + vesicles (small blisters) (+++) ; large blisters (++++)

SECONDARY OUTCOMES:
The proportion of participants who have skin irritation grade equal to or greater than two plus (++) on each assessment day (Day 3 and Day 4) | Day 3 and Day 4
  Skin irritation grade is defined as following: no reaction (-); slight erythema (+-); erythema (+); erythema + edema, papules (++); erythema + edema + papules + vesicles (small blisters) (+++) ; large blisters (++++)
The number of the maximum skin irritation score reported up to Day 4 by treatment | Up to Day 4
  Skin irritation score is defined as following: no reaction (0); slight erythema (0.5); erythema (1); erythema + edema, papules (2); erythema + edema + papules + vesicles (small blisters) (3) ; large blisters (4)
The percentage of the maximum skin irritation score reported up to Day 4 by treatment | Up to Day 4
  Skin irritation score is defined as following: no reaction (0); slight erythema (0.5); erythema (1); erythema + edema, papules (2); erythema + edema + papules + vesicles (small blisters) (3) ; large blisters (4)
The number of each skin irritation score reported by treatment on each assessment day | Day 3 and Day 4
  Skin irritation score is defined as following: no reaction (0); slight erythema (0.5); erythema (1); erythema + edema, papules (2); erythema + edema + papules + vesicles (small blisters) (3) ; large blisters (4)
The percentage of each skin irritation score reported by treatment on each assessment day | Day 3 and Day 4
  Skin irritation score is defined as following: no reaction (0); slight erythema (0.5); erythema (1); erythema + edema, papules (2); erythema + edema + papules + vesicles (small blisters) (3) ; large blisters (4)
Number of Treatment-Emergent Adverse Events (AEs) or Serious Adverse Events (SAEs) | Baseline up to Day 35
Number of Participants Discontinuation Due to AEs | Baseline up to Day 35

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Medical Corporation Heishinkai OPHAC Hospital, Osaka, Osaka, Japan

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B7931029&StudyName=A+PHASE+1%2C+SINGLE-CENTER%2C+RANDOMIZED%2C+VEHICLE+AND+WHITE+PETROLATUM+CONTROLLED%2C+EVALUATOR+BLINDED+STUDY+TO+ASSESS+THE+SKIN+IRRITATION+POTENTIAL+WITH+A+RANGE+OF+CONCENTRATIONS+OF+PF-06700841+CREAM+IN+ADULT+JAPANESE+HEALTHY+PARTICIPANTS